CLINICAL TRIAL: NCT04399811
Title: Machine Learning-Based Near-infrared Vision to Evaluate the Microcirculatory of Critical Ill Patients: A Prospective Observational Study
Brief Title: Near-infrared Vision for Microcirculatory Status
Acronym: NVIM
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: B2020-057R
Record Dates: First submitted 2020-05-16; First posted 2020-05-22 (Actual); Last update posted 2020-05-22 (Actual); Status verified 2020-05

CONDITIONS: Near-infrared Vision; Machine Learning; Microcirculatory Status

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Near-infrared Vision Photograph — The near-infrared image will be recorded (by a infrared camera connected to a laptop) for each enrolled patient

SUMMARY:
The investigators aimed to combine the image of near-infrared vision and machine learning method to evaluate the microcirculatory status of critical ill patients.

DETAILED DESCRIPTION:
The heat distribution of body is determined by the circulatory status. The investigators plan to the near-infrared vision to collect heat distribution information of limbs. Then, the machine learning method will be performed to recognize the subtle differences between images. Due to lack of golden standard of microcirculatory status, indirect parameters (such as lactate clearance, capillary refill time) and clinical outcomes will be recorded to evaluate the performance of maching learning model.

ELIGIBILITY:
Inclusion Criteria:

* Age≥18 years;
* Patients who were transfered to our ICU.

Exclusion Criteria:

* Abnormalities of lower limbs arteries

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: General critical ill patients who required evaluation of perfussion.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2020-05-17 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Hospital mortality | From date of admission to our ICU until the date of hospital discharge or date of death from any cause, whichever came first, assessed up to 2 months.
  The rate of patients who died during hospital stay.

SECONDARY OUTCOMES:
Lacteta clearance rate | When the near-infrared image is taken for a patient, the blood gas analysis will be performed immediately to get the value of lactate. After 2-hours, another blood gas analysis will be conducted to get the second value of lactete.
  The percent change of lactate between lactates measured in two time points. This parameter was usually used to guide resuscitation in septic shock.
Capillary refill time (CRT) | When the near-infrared image is taken for a patient, the capillary refill time will be measured immediately.
  A noninvasive parameter of peripheral perfusion status. CRT was measured by applying firm pressure to the ventral surface of the right index finger distal phalanx with a glass microscope slide. The pressure was increased until the skin was blank and then maintained for 10 seconds. The time for return of the normal skin color was registered with a chronometer, and a refill time greater than 3 seconds was defined as abnormal.(Hernández 2019.JAMA)

IPD SHARING:
Plan to Share IPD: No
Our institutional ethics commitee did nor approve to share data.